CLINICAL TRIAL: NCT01495000
Title: A Six-Month Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Denosumab in Indian Postmenopausal Women With Osteoporosis
Brief Title: A Study in Indian Postmenopausal Women With Osteoporosis to Evaluate the Efficacy and Safety of Denosumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114161
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2013-12

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: India; dual energy x-ray absorptiometry; bone mineral density; denosumab
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): denosumab 60mg subcutaneous injection, single dose at the start of the 6-month double-blind treatment
  Interventions: Drug: denosumab
- Arm 2 (Placebo Comparator): placebo subcutaneous injection, single dose at the start of the 6-month double-blind treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: denosumab — 60mg subcutaneous injection, single dose
  Arms: Arm 1
Drug: placebo — placebo subcutaneous injection, single dose
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine if denosumab is effective in increasing bone mineral density at the lumbar spine in Indian postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory Indian postmenopausal women with osteoporosis
* greater than 5 years postmenopausal
* aged 55 to 75 years old
* absolute bone mineral density value consistent with a T-score less than -2.5 and greater than - 4.0 at the either the lumbar spine or total hip, as measured by dual energy x-ray absorptiometry. Subjects with a T-score less than or equal to -4.0 are at very high risk for fracture and will be excluded.

Exclusion Criteria:

* previous or current metabolic bone disease, Paget's or Cushing's disease, or hyperprolactinemia
* current hypo- or hyperparathyroidism or hypo- or hyperthyroidism unless on stable thyroid replacement therapy and TSH level meets criteria
* rheumatoid arthritis
* cirrhosis of the liver or unstable liver disease or ALT or AST greater than or equal to 2.0 times the upper limit of normal, or alkaline phosphatase and bilirubin greater than or equal to 1.5 times the upper limit of normal
* medications used to treat osteoporosis, defined for type and duration of use, and including IV and oral bisphosphonates
* medications that affect bone metabolism including parathyroid hormone or derivatives; anabolic steroids or testosterone; glucocorticosteroids; systemic hormone replacement therapy; selective estrogen receptor modulators; tibolone, calcitonin, and calcitriol or vitamin D derivatives; other bone active drugs including anticonvulsives (but not benzodiazepines) and heparin; chronic systemic ketoconazole, androgens, ACTH, cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, and gonadotropin-releasing hormone agonists
* malignancy within 5 years except certain resected types
* malabsorption syndrome or gastrointestinal disorders associated with malabsorption
* abnormal calcium level
* vitamin D deficiency
* any laboratory abnormality that will prevent the subject from completing the study or interferes with interpretation of study results
* oral or dental conditions including current or past history of osteomyelitis or osteonecrosis of the jaw; active dental or jaw condition with requires oral surgery; planned invasive dental procedure; un-healed dental or oral surgery
* any disorder that compromises the ability of the subject to give written informed consent or to comply with study procedures
* any physical or psychiatric disorder that will prevent the subject from completing the study or interferes with study results
* known to have tested positive for HIV
* less than two lumbar vertebrae evaluable for DXA measurements
* height, weight, or girth that may preclude accurate DXA measurements
* drug or alcohol abuse within 12 months that interferes with understanding or completing the study
* known sensitivity to mammalian cell-derived drug products
* use of an investigational drug or device within 30 days of enrollment or currently receiving other investigational agent(s)

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- India (8):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Mangalore
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Trivandrum
  - GSK Investigational Site, Vadodra

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a Screening Phase of up to 2.5 months and a 6-month Double-blind Treatment Phase. A total of 551 participants (par.) were screened; 303 par. were screen failures, and 250 par. were randomized (2 par. were considered to be screen failures; however, these par. were randomized, 1 to each treatment group).
Groups:
- Denosumab 60 mg: Participants received denosumab 60 milligrams (mg) administered as a single subcutaneous (SC) injection at the start of the Double-blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 international units [IU]).
- Placebo: Participants received placebo administered as a single subcutaneous injection at the start of the Double-blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 IU).
Period: Overall Study
Arm/Group | Denosumab 60 mg | Placebo
Started | 124 | 126
Completed | 111 | 114
Not Completed | 13 | 12
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 60 mg | Placebo | Total
Number analyzed (Participants) | 124 | 126 | 250
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (5.10) | 62.6 (4.85) | 62.6 (4.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 126 | 250
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Central/South Asian Heritage | 124 | 126 | 250

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Bone Mineral Density at the Lumbar Spine at Month 6
Description: Bone mineral density (BMD) at the lumbar spine was measured by the dual-energy x-ray absorptiometry (DXA) scanner. The mean percent change from Baseline in BMD was calculated as: (value at Month 6 minus Baseline value) * 100 / Baseline value. Analysis was performed using an Analysis of Covariance (ANCOVA) model with terms for treatment and baseline BMD at the lumbar spine (as a continuous covariate).
Time Frame: Baseline and Month 6
Population: Intent-to-Treat Efficacy (ITTE) Population: all randomized participants who received one dose of study medication, and who had a Baseline measure and at least one post-Baseline efficacy measure during the Double-blind Treatment Phase. Only participants with BMD values at both Baseline and Month 6 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 100 | 105
percent change | 4.26 (0.413) | 1.20 (0.403)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.05, 95% CI 2-sided [1.91 to 4.19]

2. Secondary Outcome: Mean Percent Change From Baseline in BMD at the Total Hip, Femoral Neck, and Trochanter at Month 6
Description: BMD at the total hip, femoral neck, and trochanter was measured by the DXA scanner. The mean percent change from Baseline in BMD was calculated as: (value at Month 6 minus Baseline value) * 100 / Baseline value. Analysis was performed using an ANCOVA model with terms for treatment and corresponding Baseline BMD (as a continuous covariate).
Time Frame: Baseline and Month 6
Population: ITTE Population. Only participants with BMD values at both Baseline and Month 6 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 87 | 86
percent change
  Total Hip | 2.02 (0.270) | 0.32 (0.271)
  Femoral Neck | 2.69 (0.407) | 0.40 (0.409)
  Trochanter | 2.49 (0.366) | 0.69 (0.368)

3. Secondary Outcome: Median Percent Change From Baseline in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) and Serum Procollagen Type IN Propeptide (s-PINP) Markers at Months 1, 3, and 6
Description: Blood samples were collected for the measurement of s-CTx and s-PINP, which are used as biomarkers of bone resorption and formation, respectively. The median percent change from Baseline in s-CTX and s-PINP markers at Months 1, 3, and 6 was calculated as: (post-Baseline value minus Baseline value) * 100 / Baseline value.
Time Frame: Baseline; Months 1, 3, and 6
Population: ITTE Population. Only participants with s-CTX and s-PINP values at both Baseline and Months 1, 3, and 6 were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points/for different parameters, so the overall number of participants analyzed reflects the entire ITTE Population.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 121 | 123
percent change
  s-CTx, Month 1, n=112, 121 | -80.61 [-87.42 to -65.04] | -17.01 [-40.03 to 6.93]
  s-CTx, Month 3, n=107, 113 | -82.43 [-87.50 to -66.54] | -18.97 [-44.25 to 3.56]
  s-CTx, Month 6, n=105, 113 | -62.5 [-77.60 to -42.86] | -28.82 [-47.33 to -1.15]
  s-PINP, Month 1, n=110, 120 | -34.55 [-50.00 to -21.74] | -13.62 [-23.94 to -2.21]
  s-PINP, Month 3, n=107, 111 | -78.08 [-84.13 to -65.38] | -27.87 [-42.68 to -1.75]
  s-PINP, Month 6, n=104, 113 | -63.41 [-76.50 to -53.85] | -25.81 [-41.79 to 0.00]

4. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury with hyperbilirubinaemia. Medical or scientific judgment was to have been exercised in other important medical events. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From Baseline up to Month 6
Population: ITT Population: all participants who received one dose of study medication
Measure: Number; unit: participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 124 | 126
participants
  Any AE | 38 | 47
  Any SAE | 1 | 3

5. Secondary Outcome: Number of Participants With a Change From Baseline in Vital Signs of Potential Clinical Concern at Months 1, 3, and 6
Description: Vital sign values of potential clinical concern were defined as: change in heart rate >30 beats per minutes (bpm), change in systolic blood pressure (SBP) >30 millimeters of mercury (mmHg), and change in diastolic blood pressure (DBP) >20 mmHg. The number of participants with post-Baseline vital sign values of potential clinical concern who did not have values of potential clinical concern at Baseline are summarized. If the change from Baseline is a decrease greater than the threshold, it is categorized as "low." If the change from Baseline is an increase greater than the threshold, it is categorized ad "high."
Time Frame: Baseline; Months 1, 3, and 6
Population: ITT Population. Only participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points/for different parameters, so the overall number of participants analyzed reflects the entire ITT Population.
Measure: Number; unit: participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 124 | 126
participants
  DBP, Month 1: High, n=122, 125 | 1 | 2
  DBP, Month 1: Low, n=122, 125 | 1 | 4
  DBP, Month 3: High, n=117, 120 | 2 | 0
  DBP, Month 3: Low, n=117, 120 | 0 | 2
  DBP, Month 6: Low, n=111, 114 | 0 | 3
  SBP, Month 1: Low, n=122, 125 | 1 | 2
  SBP, Month 3: High, n=117, 120 | 1 | 1
  SBP, Month 3: Low, n=117, 120 | 1 | 3
  SBP, Month 6: Low, n=111, 114 | 2 | 3
  Heart Rate, Month 3: Low, n=117, 120 | 0 | 1

6. Secondary Outcome: Number of Participants With the Indicated Laboratory Parameter Values of Potential Clinical Concern at Month 6
Description: The number of participants with laboratory parameter values of potential clinical concern at Month 6 are summarized. The following are the laboratory values of potential clinical concern: alkaline phosphatase, High: >375 units/Liter (L); aspartate aminotransferase, High: >165 units/L; creatinine, High: >159 micromoles (µmol)/L; glucose, Low: <3 millimoles (mmol)/L; hematocrit, Low: <0.325; hemoglobin, Low: <91grams/L; phosphorus, High: >1.723 mmol/L; potassium, High: >6.3 mmol/L; sodium, Low: <130 mmol/L; total neutrophils, Low: <0.9 10^9 cells (GI)/L; blood urea nitrogen (BUN), High: >21mmol/L; uric acid, High: 654 µmol/L.
Time Frame: Month 6
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 124 | 126
participants
  Alkaline phosphatase: High, n=107, 114 | 0 | 1
  Aspartate aminotransferase: High, n=107, 113 | 1 | 0
  Creatinine: High, n=107, 114 | 1 | 1
  Glucose: Low, n=107, 114 | 1 | 0
  Hematocrit: Low, n=106, 111 | 1 | 1
  Hemoglobin: Low, n=106, 111 | 2 | 3
  Inorganic Phosphorus: High, n=107, 114 | 0 | 1
  Potassium: High, n=107, 113 | 1 | 0
  Sodium: Low, n=107, 114 | 0 | 1
  Total Neutrophils: Low, n=104, 107 | 0 | 2
  Urea/BUN: High, n=107, 114 | 0 | 1
  Uric Acid: High, n=107, 114 | 0 | 1

7. Secondary Outcome: Change From Baseline in Albumin/Globulin Ratio and Blood Urea Nitrogen (BUN)/Creatinine Ratio at Month 6
Description: Blood samples were collected for the measurement of albumin/globulin ratio and BUN/creatinine ratio values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 106 | 114
ratio
  Albumin/globulin ratio | 0.025 (0.1446) | 0.018 (0.1518)
  BUN/creatinine ratio | -5.896 (18.0195) | -1.860 (19.8400)

8. Secondary Outcome: Change From Baseline in Albumin, Hemoglobin, Mean Corpuscle Hemoglobin Concentration (Conc.), and Total Protein at Month 6
Description: Blood samples were collected for the measurement of albumin, hemoglobin, mean corpuscle hemoglobin concentration, and total protein values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects the entire ITT Population.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 124 | 126
grams per liter (g/L)
  Albumin, n=106, 114 | 0.689 (2.4470) | 0.746 (2.9020)
  Hemoglobin, n=106, 107 | 2.236 (6.2891) | 1.925 (8.4927)
  Mean corpuscle hemoglobin conc., n=106, 107 | 2.321 (9.8653) | 1.607 (10.0196)
  Total protein, n=106, 114 | 0.585 (3.8219) | 0.886 (4.1621)

9. Secondary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatinine Kinase, Gamma Glutamyl Transferase, and Lactate Dehydrogenase at Month 6
Description: Blood samples were collected for the measurement of alkaline phosphatase, alanine amino transferase, aspartate amino transferase, creatinine kinase, gamma glutamyl transferase, and lactate dehydrogenase values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 124 | 126
International units per liter (IU/L)
  Alkaline phosphatase, n=106, 114 | -18.179 (25.0207) | -3.684 (41.4420)
  Alanine amino transferase, n=106, 114 | 2.481 (10.2421) | 0.035 (15.6640)
  Aspartate amino transferase, 106, 113 | 2.755 (10.9465) | -0.965 (16.9226)
  Creatinine kinase, n=106, 114 | 6.170 (51.2968) | 11.175 (63.0331)
  Gamma glutamyl transferase, n=106, 114 | 2.915 (12.8346) | -0.754 (13.8433)
  Lactate dehydrogenase, n=106, 113 | 2.764 (25.2811) | 0.434 (36.7389)

10. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Segmented Neutrophils, Total Neutrophils, Platelet Count, and White Blood Cell Count Month 6
Description: Blood samples were collected for the measurement of basophil, eosinophil, lymphocyte, monocyte, segmented neutrophil, total neutrophil, platelet count, and white blood cell count values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 124 | 126
10^9 cells per liter (GI/L)
  Basophils, n=104, 103 | 0.001 (0.0221) | -0.001 (0.0262)
  Eosinophils, n=104, 103 | -0.076 (0.2794) | -0.001 (0.3414)
  Lymphocytes, n=104, 103 | -0.065 (0.6044) | -0.056 (0.7476)
  Monocytes, n=104, 103 | 0.000 (0.1204) | 0.032 (0.1727)
  Segmented neutrophils, n=104, 103 | -0.290 (1.6142) | -0.129 (1.7405)
  Total neutrophils, n=104, 103 | -0.297 (1.6099) | -0.135 (1.7343)
  Platelet count, n=103, 105 | 3.117 (38.5322) | 7.533 (36.5761)
  White blood cell count, n=104, 103 | -0.436 (1.6614) | -0.160 (1.7629)

11. Secondary Outcome: Change From Baseline in Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, Creatinine, and Uric Acid at Month 6
Description: Blood samples were collected for the measurement of direct bilirubin, indirect bilirubin, total bilirubin, creatinine, and uric acid values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micromoles per liter (UMOL/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 124 | 126
micromoles per liter (UMOL/L)
  Direct bilirubin, n=105, 112 | 0.152 (1.1667) | 0.089 (1.2122)
  Indirect bilirubin, n=105, 112 | 0.210 (2.7305) | -0.054 (2.2050)
  Total bilirubin, n=106, 114 | 0.358 (2.8659) | 0.000 (2.2102)
  Creatinine, n=106, 114 | 2.337 (11.8458) | 3.041 (13.1471)
  Uric acid, n=106, 114 | -2.642 (60.6677) | -6.316 (61.9058)

12. Secondary Outcome: Change From Baseline in Calcium Corrected, Calcium, Chloride, Glucose, Potassium, Magnesium, Sodium, Phosphorus Inorganic, Triglycerides, Urea/BUN, and Very Low-density Lipoproteins (VLDL) Cholesterol Calculation at Month 6
Description: Blood samples were collected for the measurement of calcium corrected, calcium, chloride, glucose, potassium, magnesium, sodium, phosphorus inorganic, triglyceride, urea/BUN, and VLDL cholesterol calculation values. Change from Baseline was calcualted as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimoles per liter (MMOL/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 124 | 126
millimoles per liter (MMOL/L)
  Calcium corrected, n=12, 24 | 0.015 (0.0573) | 0.008 (0.0755)
  Calcium, n=106, 113 | 0.012 (0.1194) | 0.033 (0.1069)
  Chloride, n=106, 114 | -0.802 (3.0376) | -0.895 (3.0552)
  Glucose, n=106, 113 | -0.571 (2.2401) | -0.303 (2.6346)
  Potassium, n=106, 113 | 0.140 (0.4581) | 0.158 (0.4118)
  Magnesium, n=106, 114 | 0.009 (0.0718) | 0.009 (0.0614)
  Sodium, n=106, 114 | -0.472 (2.2979) | -0.395 (2.5921)
  Phosphorus inorganic, n=106, 114 | -0.052 (0.2047) | -0.012 (0.1674)
  Triglycerides, n=106, 114 | -0.305 (0.7413) | -0.263 (0.8433)
  Urea/BUN, n=106, 114 | -0.283 (1.1423) | 0.114 (2.2032)
  VLDL cholesterol calculation, n=103, 109 | -0.131 (0.3178) | -0.105 (0.3504)

13. Secondary Outcome: Change From Baseline in Hematocrit at Month 6
Description: Blood samples were collected for the measurement of hematocrit values. Change from Baseline was calculated as the Month 6 value minuse the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: proportion of RBCs in blood
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 106 | 107
proportion of RBCs in blood | 0.004 (0.0204) | 0.004 (0.0264)

14. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin at Month 6
Description: Blood samples were collected for the measurement of hemoglobin values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 106 | 107
picograms | 0.407 (0.8613) | 0.260 (1.2787)

15. Secondary Outcome: Change From Baseline in Mean Corpuscular Volume at Month 6
Description: Blood samples were collected for the measurement of mean corpuscular volume values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 106 | 107
femtoliters | 0.623 (2.9775) | 0.327 (3.5309)

16. Secondary Outcome: Change From Baseline in Red Blood Cell Count at Month 6
Description: Blood samples were collected for the measurement of red blood cell count values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 106 | 107
10^12 cells per liter (TI/L) | 0.016 (0.2575) | 0.034 (0.3034)

17. Secondary Outcome: Change From Baseline in Red Cell Distribution Width at Month 6
Description: Blood samples were collected for the measurement of red cell distribution width values. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 106 | 107
percentage | 0.065 (1.2126) | -0.121 (1.2735)

18. Secondary Outcome: Number of Participants With Positive and Negative Results for Anti-body Formation to Denosumab at Month 6
Description: The number of participants with positive and negative results for both neutralizing antibodies to denosumab and for binding antibodies to denosumab at Month 6 are summarized.
Time Frame: Month 6
Population: ITT Population. Only participants available at the specified time point were analyzed.
Measure: Number; unit: participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 110 | 114
participants
  Neutralizing antibodies, n=0, 0 | NA — Participants were only to have been analyzed for neutralizing antibodies in the event that they were positive for binding antibodies. Because no participants were positive for binding antibodies, no analysis was conducted for neutralizing antibodies. | NA — Participants were only to have been analyzed for neutralizing antibodies in the event that they were positive for binding antibodies. Because no participants were positive for binding antibodies, no analysis was conducted for neutralizing antibodies.
  Binding antibodies, Positive, n=110, 114 | 0 | 0
  Binding antibodies, Negative, n=110, 114 | 110 | 114

ADVERSE EVENTS:
Time Frame: SAEs (serious adverse events) and non-serious AEs were collected from the start of study medication through the study period (6-month post-dose) (up to Study Week 43).
Description: AEs and SAEs were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who received one dose of study medication.
Arm/Group | Denosumab 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/124 | 3/126
Other Adverse Events (participants affected / at risk) | 8/124 | 3/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 60 mg (N=124) | Placebo (N=126)
Hypotension (Vascular disorders) | 0 | 1
Varicose vein ruptured (Vascular disorders) | 0 | 1
Cataract nuclear (Eye disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 60 mg (N=124) | Placebo (N=126)
Upper respiratory tract infection (Infections and infestations) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.